CLINICAL TRIAL: NCT06821386
Title: N-Care Project: Enhancing Asian-Pacific Collaboration
Acronym: N-Care project
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202412119RINA
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Whole Genome Sequencing; Genetic Disease; Critical Care, Intensive Care; Nanopore Sequencing
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted the DNA from 3-5cc whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Genetic study with nanopore sequencing — The study targets critically ill children under 18 months of age, employing third-generation genome sequencing technology to complete long-read sequencing within 8-11 days, analyzing single nucleotide variants, small insertions/deletions, and structural variations. Through this research, we aim to enhance diagnostic accuracy, enabling ICUs to provide personalized and precision care and treatment based on genetic information, thereby ensuring a greater level of health security for these children. We only draw 3-5cc whole blood once for exam.

SUMMARY:
Through Asian-Pacific multinational collaboration, we aim to utilize third-generation genome sequencing to rapidly diagnose genetic diseases in critically ill infants and young children, achieving the goal of early diagnosis for targeted treatment.

DETAILED DESCRIPTION:
A group of individuals with specific characteristics was selected. Genetic studies were arranged for participants who provided their consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age: infant/newborn less than 18 months
2. Admitted to intensive care unit
3. At least one of the following conditions A. Specific anomaly highly suggestive of a genetic etiology

   * Multiple birth defects
   * Single major malformation that required intervention (surgery or medication)
   * Significantly abnormal EKG
   * Significant hypotonia

B. Children with high-risk stratification on assessment of a Brief Resolved Unexplained Event (BRUE) with any of the following:

* Recurrent severe infection events
* Recurrent or prolonged seizures
* Unexplained cardiopulmonary resuscitation (CPR)
* Suspect inborn error of metabolism

Exclusion Criteria:

1. Infants with a definitive non-genetic diagnosis: ex as below A. An infection with normal response to therapy B. Isolated prematurity C. Transient hypoglycemia D. Isolated unconjugated hyperbilirubinemia E. Isolated Transient Neonatal Tachypnea F. Those where the clinical course can be explained without genetic testing
2. Confirmed genetic diagnosis explains illness
3. Lack of consent: Families who do not consent to genetic testing or data sharing.
4. Infants without sufficient DNA sample quality/quantity: Where the quality or quantity of the DNA sample is inadequate for sequencing.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants or newborns under 18 months of age admitted to the ICU with a high suspicion of a genetic disease.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive yield rate | 9 days after enrollment
  The percentage of individuals who test positive among the long-read sequencing exam

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan